CLINICAL TRIAL: NCT07082322
Title: European Prospective Bloodstream Infection Cohort
Acronym: EPIC-BSI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Philipp Mathe, Prof. Siegbert Rieg/Dr. Philipp Mathé, University Hospital Freiburg
Other Study IDs: 24-1521-S1
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Bloodstream Infection
Keywords: Registry; Therapeutical management
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Microbiological isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EPIC BSI Registry: Registry of bloodstream infection patients from microbiological databases
- EPIC BSI Diagnostics: Repeated survey of participating centers regarding their diagnostic standard of care
- EPIC BSI Management: Registry of bloodstream infection patients with focus on clinical course and management

SUMMARY:
Background:

Bloodstream infections (BSIs) and sepsis continue to pose significant public health challenges, contributing to high morbidity and mortality worldwide. According to the Global Burden of Diseases Study, BSIs and sepsis are associated with approximately 20% of global deaths. However, the clinical characteristics of BSIs have evolved over recent years, showing significant variability across different countries and continents. The diversity in management standards across regions further complicates the generalization and transferability of research findings. Despite the critical need for comprehensive data, BSI research in Europe remains fragmented, often limited to national-level studies.

Project Aim:

The EPIC-BSI project aims to address these challenges by establishing a multinational, collaborative bloodstream infection cohort across Europe and globally. The primary objectives are to:

* Integrate national BSI research into a cohesive multinational cohort that enable large-scale comparative research by standardizing BSI incidence data, diagnostic and therapeutic approaches, and patient outcomes across European countries and beyond.
* Monitor shifts in BSI characteristics, including the emergence of multi-drug resistant organisms, and changes in risk groups, diagnostics, and therapies.
* Create a foundation for future studies and collaborations, such as integrating BSI data with international antibiotic usage, population data, health policy data, or by biobanking blood-borne pathogens for sequencing.

The study is divided into three arms focusing on BSI epidemiology (EPIC-BSI registry), diagnostics (EPIC-BSI Diagnostic Study) and management (EPIC-BSI Management study). The EPIC-BSI Management study is partitioned in different levels of data contribution to reduce barriers for centres and enable broad participation.

Specific Objectives and Endpoints:

EPIC-BSI Registry:

* Primary aim/endpoint: Establish an international prospective BSI cohort with anonymized inclusion of all BSI cases from participating centres allowing estimation of BSI incidence by pathogen in the participating centres.
* Secondary aims/endpoints:

  * Analyse the incidence of BSIs across different settings and countries.
  * Monitor changes in patient demographics (age, gender) and acquisition modes.
  * Track shifts in antimicrobial resistance patterns.
  * Review effects of infection control practices on MDRO-BSI frequency

EPIC-BSI Diagnostic Study:

* Primary aim/endpoint: Biannual evaluation of diagnostic procedures and standards regarding BSI at participating centres
* Secondary aims/endpoints:

  * Assess the availability and use of (new) clinical and microbiological diagnostics.
  * Identify gaps in diagnostic practices and time lags between scientific evidence, guideline publication and clinical implementation of new diagnostic utilities.

EPIC-BSI Management Study:

* Primary aim/endpoint: Analyse clinical data from BSI cases to evaluate management practices regarding the effect on in-hospital mortality and outcome on day 90 after onset incl. patient-reported outcomes (Desirability-of-outcome-ranking (DOOR) or health-related quality of life metrics)
* Secondary aims/endpoints:

  * Identify differences in clinical management across countries and hospital types.
  * Analyse the impact of antimicrobial resistance patterns on clinical outcomes.
  * Evaluate the effectiveness of different established therapeutic regimens.

ELIGIBILITY:
Inclusion Criteria:

* EPIC-BSI Registry: Positive blood cultures result. For each patient only the first positive blood culture result during 90 days would be counted.
* EPIC-BSI Diagnostic study: Centre recruiting for the EPIC study with access to microbiological and clinical data.
* EPIC-BSI Management study - Regular dataset: First two BSI cases per month of (at least two or three) target pathogens (S. aureus, E. faecalis/E. faecium, E. coli, Klebsiella spp., P. aeruginosa, A. baumanii, Streptococcus spp.)

Exclusion Criteria:

* EPIC-BSI Registry: Non-comprehensive documentation and reporting of BSI cases, Age < 18 years
* EPIC-BSI Diagnostic Study: EPIC BSI centre does not participate in the EPIC BSI Diagnostic Study arm
* EPIC-BSI Management Study: Non-comprehensive documentation and reporting of BSI cases; Age < 18 years; For Follow-up part: Patient with dementia or other progressed neurological or vigilance disorder without contact details of legal representative, which makes follow-up unfeasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are hospitalised with a blood culture-detected bloodstream infection are eligible for inclusion into this study.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of bloodstream infections | 5 years, analysed aggregated by year
  Incidence of bloodstream infection patients stratified by pathogen
In hospital mortality | Hospital stay after infection onset until discharge, an average of 3 weeks
  Fraction of patients that died during hospital stay

SECONDARY OUTCOMES:
Patient-reported health quality | Day 90 after onset
  Patient reported health-related quality of life at day 90 measured by the EQ-5D-5L (European Quality of Life 5 Dimensions 5 Level Version) questionaire ranging between 0 (very bad) to very good (1)
Mortality at day 90 | Day 90
  Overall and infection-attributable mortality at day 90 after onset

CONTACTS AND LOCATIONS:
Overall Officials: Siegbert Rieg, Prof. Dr., Principal Investigator — University Hospital Freiburg; Philipp Mathé, Dr., Principal Investigator — University Hospital Freiburg
Locations (1):
- University Hospital Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Yes
All data analyses and publications are carried out with anonymized data, so that no conclusions can be drawn about the respective patients. At the end of the study, the anonymised data will be saved in a corresponding database for fur- ther scientific use by other research groups upon reasonable request.